CLINICAL TRIAL: NCT01388153
Title: Randomized, Non-blinded, 3-fold Crossover Study to Investigate the Bioequivalence Between Glucobay ODT Taken Without and With Water and the Glucobay Standard Tablet Following Single Oral Dosing in Healthy Male Subjects
Brief Title: A 3-fold Crossover Bioequivalence Study Between Glucobay Orally Disintegrating Tablet (ODT) and Glucobay Standard Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer Healthcare AG
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 15624; 2011-000904-17 (EudraCT Number)
Record Dates: First submitted 2011-07-04; First posted 2011-07-06 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Bioequivalence, acarbose, ODT
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Acarbose (Glucobay ODT, BAYG5421)
- Arm 2 (Experimental)
  Interventions: Drug: Acarbose (Glucobay ODT, BAYG5421)
- Arm 3 (Active Comparator)
  Interventions: Drug: Acarbose (Glucobay, BAYG5421)

INTERVENTIONS:
Drug: Acarbose (Glucobay ODT, BAYG5421) — Day 1: oral sucrose load (75 g sucrose dissolved in 225 mL water) without Glucobay ODT; Day 2: oral sucrose load plus Glucobay ODT taken without water
  Arms: Arm 1
Drug: Acarbose (Glucobay ODT, BAYG5421) — Day 1: oral sucrose load (75 g sucrose dissolved in 225 mL water) without Glucobay ODT; Day 2: oral sucrose load plus Glucobay ODT taken with water
  Arms: Arm 2
Drug: Acarbose (Glucobay, BAYG5421) — Day 1: oral sucrose load (75 g sucrose dissolved in 225 mL water) without Glucobay standard tablet; Day 2: oral sucrose load plus Glucobay standard tablet taken with water
  Arms: Arm 3

SUMMARY:
To establish the bioequivalence between Glucobay ODT (Orally Disintegrating Tablet) taken without or with water and the Glucobay standard tablet taken with water

ELIGIBILITY:
Inclusion Criteria:

* The informed consent must be signed before any study specific tests or procedures are done
* Healthy male subject
* Age: 18 to 45 years (inclusive) at the first screening examination / visit
* Ethnicity: White
* Body mass index (BMI): above/equal 18 and below/equal 28 kg / m²
* Confirmation of the subject's health insurance coverage prior to the first screening examination / visit
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Subjects with a medical disorder, condition or history of such that would impair the subject's ability to participate or complete this study in the opinion of the investigator or the sponsor
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Chronic intestinal disorders associated with distinct disturbances of digestion and absorption
* States which may deteriorate as a result of increased gas formation in the intestine (e.g. Roemheld´s syndrome, major hernias, intestinal obstructions, intestinal ulcers, Crohn´s disease, ulcerative colitis, malabsorptions)
* Fasting blood glucose level outside normal range
* Impaired glucose tolerance in glucose tolerance test

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Difference of postprandial maximum concentration (Cmax) of blood glucose following sucrose load without (Day 1) and with Glucobay (Day 2) | within 4 hours after sucrose load
Difference of postprandial Area under curve from 0 to 4 hours (AUC(0-4)) of blood glucose following sucrose load without (Day 1) and with Glucobay (Day 2) | within 4 hours after sucrose load

SECONDARY OUTCOMES:
Time to reach maximum drug concentration in plasma after single dose (tmax) of blood glucose following sucrose load without (Day 1) and with Glucobay (Day 2) | within 4 hours after sucrose load
Difference of postprandial Cmax of serum insulin following sucrose load without (Day 1) and with Glucobay (Day 2) | within 4 hours after sucrose load
Difference of postprandial AUC(0-4) of serum insulin following sucrose load without (Day 1) and with Glucobay (Day 2) | within 4 hours after sucrose load
Tmax of serum insulin following sucrose load without (Day 1) and with Glucobay (Day 2) | within 4 hours after sucrose load

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mönchengladbach, North Rhine-Westphalia, Germany